CLINICAL TRIAL: NCT03685812
Title: Validity and Reliability of Autocad Software Assessment of Joint Position Sense in Patellofemoral Pain Syndrome
Brief Title: Validity and Reliability of Autocad Software Assessment of JPS in PFPS
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karima Abdelaty Hassan, principal investigator, Cairo University
Other Study IDs: patellofemoral pain syndrome
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral Pain Syndrome; Autocad software; position sense; validity; reliability
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with patellofemoral pain syndrome , Auto Cad software: Patients referred with a confirmed diagnosis of patellofemoral pain syndrome, with a visual analogue scale of more than 3. Anterior or retropatellar knee pain from at least 2 of the following Activities : (1) prolonged sitting; (2) stair climbing; (3) squatting; (4) running; (5) kneeling; and (6) hopping/jumping.
  Interventions: Diagnostic Test: Autocad software

INTERVENTIONS:
Diagnostic Test: Autocad software — The participants will be prepared for image-capture data collection by putting four squared markers on leg and thigh.Each subject will extend his/her leg and make two angles from the resting position (90º) to the full extension, photos will be taken. The tested leg passively moved by the researcher through 20° to 60° of knee extension, the participant will be instructed to actively move that leg to the target angle and hold it in this position another photograph will be taken. The angles will be measured using the AutoCAD software. Knee JPS measurements will also be collected using an IKD by same steps
  Other Names: Isokinetic system

SUMMARY:
The overall aim of the study is to assess the reliability and validity of Autocad software to measure JPS in PFPS, especially:

1. To assess the intra-tester and between day reliability of measurement of JPS using Autocad software.
2. To assess the validity of these measurements against those found during an IKD.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is a common painful musculoskeletal condition that affects physically active young adults and adolescents.

Joint position sense (JPS) is considered as a component of proprioception as it provides the clinician with information regarding the accuracy of movement as well as its relationship with movement performance and injuries. Therefore researchers use advanced instruments as 3 D video systems and isokinetic dynamometer. Since these instruments are less portable and expensive, therefore researchers used another method to evaluate JPS using high precision software using video analysis and markers in the joints. Unfortunately, video analysis requires difficult and time-consuming tasks and that this slow the evaluation process.

Although immediate feedback could help physiotherapists and athletic trainers to monitor athletes and make decisions during the training session and the rehabilitation process, such immediacy is not available for proprioceptive tests in field situations. Autocad software is available and inexpensive and provides immediate feedback

ELIGIBILITY:
inclusion criteria:

1. Anterior or retropatellar knee pain from at least 2 of the following Activities : (1) prolonged sitting; (2) stair climbing; (3) squatting; (4) running; (5) kneeling; (6) hopping/jumping; (7) kneel sitting
2. Insidious onset of symptoms unrelated to a traumatic incident.
3. Age of the subject 18-35 years to limit the possibility that PFPS over age 35 may have been complicated by arthritic changes, and also the subjects should have closed epiphyseal growth plates.
4. Patient with chronic PFPS (pain > 3 months)

Exclusion Criteria:

1. Meniscal or other intraarticular pathologic conditions; cruciate or collateral ligament involvement.
2. A history of traumatic patellar subluxation or dislocation.
3. Previous surgery in the knee, ankle and hip joints.
4. Knee, ankle and hip joints osteoarthritis.
5. athletes weren't included.

   -

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: thirty-eight patients(males and females) with PFPS will be recruited from the outpatient clinic of the faculties of Physical Therapy, Cairo University, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Concurrent validity of Autocad software | one day
  correlation between absolute angular error of Autocad software and isokinetic system

SECONDARY OUTCOMES:
Intrarater reliability of | 48 hours
  same investigator will repeat joint positsion sense by Autocad software

CONTACTS AND LOCATIONS:
Overall Officials: karima A Hassan, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akseki D, Akkaya G, Erduran M, Pinar H. [Proprioception of the knee joint in patellofemoral pain syndrome]. Acta Orthop Traumatol Turc. 2008 Nov-Dec;42(5):316-21. doi: 10.3944/aott.2008.316. Turkish. PMID 19158451
- [Background] Baker V, Bennell K, Stillman B, Cowan S, Crossley K. Abnormal knee joint position sense in individuals with patellofemoral pain syndrome. J Orthop Res. 2002 Mar;20(2):208-14. doi: 10.1016/S0736-0266(01)00106-1. PMID 11918299
- [Background] Drouin JM, Valovich-mcLeod TC, Shultz SJ, Gansneder BM, Perrin DH. Reliability and validity of the Biodex system 3 pro isokinetic dynamometer velocity, torque and position measurements. Eur J Appl Physiol. 2004 Jan;91(1):22-9. doi: 10.1007/s00421-003-0933-0. Epub 2003 Sep 24. PMID 14508689
- [Background] Relph N, Herrington L. Criterion-related validity of knee joint-position-sense measurement using image capture and isokinetic dynamometry. J Sport Rehabil. 2015 Jan 13;24(1):2013-0119. doi: 10.1123/jsr.2013-0119. Print 2015 Feb 1. PMID 25310567
- [Background] Mir SM, Hadian MR, Talebian S, Nasseri N. Functional assessment of knee joint position sense following anterior cruciate ligament reconstruction. Br J Sports Med. 2008 Apr;42(4):300-3. doi: 10.1136/bjsm.2007.044875. PMID 18390774
- [Background] Bolgla LA, Boling MC. An update for the conservative management of patellofemoral pain syndrome: a systematic review of the literature from 2000 to 2010. Int J Sports Phys Ther. 2011 Jun;6(2):112-25. PMID 21713229